CLINICAL TRIAL: NCT00000534
Title: Calcium for Pre-Eclampsia Prevention (CPEP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: 77
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Diseases; Eclampsia; Heart Diseases; HELLP Syndrome; Hypertension; Pre-Eclampsia; Pregnancy Toxemias; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Eclampsia; Heart Diseases; HELLP Syndrome; Hypertension; Pre-Eclampsia; Vascular Diseases | interventions — Calcium; Dietary Supplements

INTERVENTIONS:
Drug: calcium
Behavioral: dietary supplements

SUMMARY:
To evaluate the efficacy of 2 grams per day of oral calcium supplementation in reducing the combined incidence of hypertensive disorders of pregnancy: pre-eclampsia, eclampsia, and the HELLP Syndrome (hypertension, thrombocytopenia, hemolysis, and abnormal liver function). The National Institute of Child Health and Human Development (NICHD) initiated the trial in 1991, with joint funding provided by the National Heart, Lung, and Blood Institute in fiscal years 1992, 1993, and 1995.

DETAILED DESCRIPTION:
BACKGROUND:

A considerable body of data has associated lower blood pressures with higher levels of dietary calcium. Epidemiologic studies, laboratory evaluations, and clinical trials have also indicated that the incidence of hypertensive disorders of pregnancy is affected similarly by calcium intake. A meta-analysis of five controlled clinical trials of calcium supplementation in pregnancy suggested a significant reduction in proteinuric pre-eclampsia of 46 percent. Several of the trials, however, suffered from 'pitfalls' in the diagnosis of pre-eclampsia, including lack of blinding, uncertain definition of endpoints, and unknown techniques of measurement. Most trials have not assessed the role of dietary nutrients or the possibility that a subgroup with low baseline urinary calcium may benefit most from calcium supplementation. In no trial has the potential for increased risk of kidney stones in the treatment group been examined systematically. Moreover, the daily schedule for administration of calcium, has generally not been reported. There was a great need, therefore, to evaluate the efficacy of calcium supplementation for the prevention of pre-eclampsia in a large multicenter controlled clinical trial. The trial considered the role of dietary nutrients, establish whether treatment is beneficial only for those with low baseline urinary calcium, conduct systematic surveillance for urolithiasis, and employ standardized terminology, techniques of measurement, and diagnostic criteria. The NHLBI provided funding to NICHD for three years by means of an Intraagency Agreement (Y01HC20154).

DESIGN NARRATIVE:

Randomized, double-blind, multicenter. Healthy nulliparous patients were randomly assigned to receive either 2 grams of supplemental calcium daily ((n = 2,295) or placebo (n = 2,294) in a double-blind study. Study tablets were administered beginning from 13 to 21 completed weeks of gestation and continued until the termination of pregnancy. Eligible patients entered a run-in period of 6 to 14 days to exclude highly noncompliant subjects. During the run-in, obstetrical ultrasound was performed if it had not been obtained previously, and blood was drawn for serum calcium and creatinine. Follow-up visits were scheduled every four weeks through the 29th week of gestation, then every two weeks through the 35th week, and weekly thereafter. Blood pressure and urine-protein were obtained at each clinic visit, during labor and delivery, and during the first 24 hours postpartum. Primary endpoints included pregnancy-associated hypertension, pregnancy-associated proteinuria, pre-eclampsia, eclampsia, or hypertension. Other endpoints included placental abruption, cerebral hemorrhage or thrombosis, elevated liver enzymes, acute renal failure, and disseminated intravascular coagulation. Surveillance was conducted for renal calculi. Recruitment began in May 1992 and ended in March 1995. Follow-up was completed in October of 1995. Data analysis continued through March 2000 under the NICHD contract N01HD13121.

ELIGIBILITY:
Nulliparous, normotensive, pregnant women.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1991-03; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Catalano — Case Western Reserve University; Luis Curet — University of New Mexico; John Hauth — University of Alabama at Birmingham; Cynthia Morris — Oregon Health and Science University; Baha Sibai — University of Tennessee

REFERENCES:
- [Background] Levine RJ, Esterlitz JR, Raymond EG, DerSimonian R, Hauth JC, Ben Curet L, Sibai BM, Catalano PM, Morris CD, Clemens JD, Ewell MG, Friedman SA, Goldenberg RL, Jacobson SL, Joffe GM, Klebanoff MA, Petrulis AS, Rigau-Perez JG. Trial of Calcium for Preeclampsia Prevention (CPEP): rationale, design, and methods. Control Clin Trials. 1996 Oct;17(5):442-69. doi: 10.1016/s0197-2456(96)00106-7. PMID 8932976
- [Background] Sibai BM, Ewell M, Levine RJ, Klebanoff MA, Esterlitz J, Catalano PM, Goldenberg RL, Joffe G. Risk factors associated with preeclampsia in healthy nulliparous women. The Calcium for Preeclampsia Prevention (CPEP) Study Group. Am J Obstet Gynecol. 1997 Nov;177(5):1003-10. doi: 10.1016/s0002-9378(97)70004-8. PMID 9396883
- [Background] Mills JL, DerSimonian R, Raymond E, Morrow JD, Roberts LJ 2nd, Clemens JD, Hauth JC, Catalano P, Sibai B, Curet LB, Levine RJ. Prostacyclin and thromboxane changes predating clinical onset of preeclampsia: a multicenter prospective study. JAMA. 1999 Jul 28;282(4):356-62. doi: 10.1001/jama.282.4.356. PMID 10432033
- [Background] Joffe GM, Esterlitz JR, Levine RJ, Clemens JD, Ewell MG, Sibai BM, Catalano PM. The relationship between abnormal glucose tolerance and hypertensive disorders of pregnancy in healthy nulliparous women. Calcium for Preeclampsia Prevention (CPEP) Study Group. Am J Obstet Gynecol. 1998 Oct;179(4):1032-7. doi: 10.1016/s0002-9378(98)70210-8. PMID 9790393
- [Background] Levine RJ, Hauth JC, Curet LB, Sibai BM, Catalano PM, Morris CD, DerSimonian R, Esterlitz JR, Raymond EG, Bild DE, Clemens JD, Cutler JA. Trial of calcium to prevent preeclampsia. N Engl J Med. 1997 Jul 10;337(2):69-76. doi: 10.1056/NEJM199707103370201. PMID 9211675